CLINICAL TRIAL: NCT04505956
Title: Prospective Randomized Double Blind Clinical Trial to Compare Holmium Laser Lithotripsy With and Without Moses Laser Technology for the Ureteroscopic Treatment of Nephrolithiasis
Brief Title: A Comparison of Ureteroscopic Treatment of Nephrolithiasis With and Without Moses Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Nicole L. Miller, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Moses Ureteroscopy RCT
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Nephrolithiasis
Keywords: Ureteroscopy; Nephrolithiasis; Kidney Stone; Lithotripsy; Holmium; Moses
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Moses Laser Lithotripsy (Experimental): Patients will have flexible URS performed in standard fashion, without deviation from the standard of care. Laser settings will be at the surgeons' discretion but will be within the range identified as standard for dusting technique using Moses laser technology.
  Interventions: Device: Holmium laser lithotripsy with Moses Technology
- Standard Laser Lithotripsy (Active Comparator): Patients will have flexible URS performed in standard fashion, without deviation from the standard of care. Laser settings will be at the surgeons' discretion but will be within the range identified as standard for dusting technique (between 0.2-0.5 J and 40-80 Hz). The short pulse setting will be utilized for non-Moses settings.
  Interventions: Device: Holmium laser lithotripsy without Moses Technology

INTERVENTIONS:
Device: Holmium laser lithotripsy with Moses Technology — Holmium laser energy will be delivered for the ureteroscopic fragmenting of kidney stones. Energy will be generated by the commercial available, FDA approved Lumenis PulseTM P120H laser system and Moses laser fiber. Renal stones will be fragmented using a dusting technique. Moses laser settings will be turned on.
  Other Names: Moses Laser Lithotripsy
  Arms: Moses Laser Lithotripsy
Device: Holmium laser lithotripsy without Moses Technology — Holmium laser energy will be delivered for the ureteroscopic fragmenting of kidney stones. Energy will be generated by the commercial available, FDA approved Lumenis PulseTM P120H laser system and Moses laser fiber. Renal stones will be fragmented using a dusting technique. Moses laser settings will be turned off.
  Other Names: Standard Laser Lithotripsy
  Arms: Standard Laser Lithotripsy

SUMMARY:
Flexible ureteroscopy is characterized as first-line therapy for the treatment of renal stones < 2 cm in size. This involves passing a flexible endoscope into the renal pelvis through the urethra, bladder and ureter in a retrograde fashion. Holmium: YAG laser remains the preferred energy modality to subsequently break stones of this size into fragments small enough to remove or pass spontaneously through the ureter. Advances in the understanding of laser energy delivery have led to the recent commercialization of the "Moses Effect" - the creation of vapor bubbles/cavities between the laser fiber tip and the target through which laser energy can more efficiently travel. Lumenis was the first to optimize this laser phenomenon and market it as "Moses Technology" in their Lumenis Pulse P120H laser system. This system is already FDA approved through the 510K pathway and is commercially available. The purpose of this study is to evaluate the potential of Moses laser technology to reduce operative time compared to non-Moses settings for ureteroscopic treatment of nephrolithiasis.

DETAILED DESCRIPTION:
There is ongoing debate on the optimal means of laser stone fragmentation, and Moses technology is the latest advancement to raise questions regarding clinical utility. Initial preclinical studies demonstrated significantly reduced stone retropulsion and higher stone ablation volume with Moses technology, leading to the conclusion that the system allows more efficient laser lithotripsy. Human studies also showed that laser lithotripsy with Moses technology utilized laser energy in less time for stone fragmentation: 10.0 (2.6-15.0) min without vs 6.0 (2.8-13.0) min with Moses technology.

Others have evaluated the cost effectiveness of Moses technology in their own cohort of 40 patients who underwent standard laser lithotripsy by comparing a 35% projected decrease in procedure time against the cost of the Moses laser fiber and machine. Mean stone size was 10.2 mm in this group of patients, and mean lasing time was 3.0 minutes. While a significant positive association was seen between stone size and laser time, cost analysis failed to show a benefit in using Moses technology across sizes.

To date, there are limited clinical data obtained through rigorous study methodology. In addition, knowledge gaps remain regarding the effect of Moses technology on other clinically meaningful outcomes such as stone-free rate. Therefore, the investigators propose a multi-center, prospective, randomized, double blind clinical trial to further assess the effect of Moses technology for lithotripsy. The investigators aim to study a broader range of outcomes which will be facilitated by being the largest study to date. The investigators also aim to study novel outcomes such as grading retropulsion and visibility by independent blinded review as well as effects of Moses technology on independently reducing surgeon burnout. Indeed, a randomized, double blind clinical trial evaluating Moses technology in 66 patients undergoing ureteroscopy was presented as a 2018 European Association of Urology abstract. While this single center study demonstrated safety and reduced fragmentation time as well as procedure time using Moses technology, it did not show a significant difference in stone-free rates. This study is also yet to be published as a manuscript.

ELIGIBILITY:
Inclusion Criteria:

* Solitary renal stone 8 to 20 mm in size or in the case of multiple stones the conglomerate diameter (additive maximal diameter of all stones on axial imaging of computed tomography) of 8-20 mm is required
* Must be a suitable operative candidate for flexible ureteroscopy per urologic guidelines
* Must be 18 years or older
* Must be able to give consent

Exclusion Criteria:

* Concomitant stones in the ureter
* Prior ipsilateral upper urinary tract reconstructive procedures or history of ipsilateral ureteral stricture
* Prior radiotherapy to the abdomen or pelvis
* Neurogenic bladder or spinal cord injury
* Pregnancy
* Untreated UTI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole L Miller, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (6):
- United States (6):
  - Mayo Clinic, Phoenix, Arizona
  - University of California San Diego, San Diego, California
  - Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART II. J Urol. 2016 Oct;196(4):1161-9. doi: 10.1016/j.juro.2016.05.091. Epub 2016 May 27. PMID 27238615
- [Background] Turk C, Petrik A, Sarica K, Seitz C, Skolarikos A, Straub M, Knoll T. EAU Guidelines on Interventional Treatment for Urolithiasis. Eur Urol. 2016 Mar;69(3):475-82. doi: 10.1016/j.eururo.2015.07.041. Epub 2015 Sep 4. PMID 26344917
- [Background] Ventimiglia E, Traxer O. What Is Moses Effect: A Historical Perspective. J Endourol. 2019 May;33(5):353-357. doi: 10.1089/end.2019.0012. PMID 30892062
- [Background] Law KE, Lowndes BR, Kelley SR, Blocker RC, Larson DW, Hallbeck MS, Nelson H. NASA-Task Load Index Differentiates Surgical Approach: Opportunities for Improvement in Colon and Rectal Surgery. Ann Surg. 2020 May;271(5):906-912. doi: 10.1097/SLA.0000000000003173. PMID 30614878
- [Background] Dias RD, Ngo-Howard MC, Boskovski MT, Zenati MA, Yule SJ. Systematic review of measurement tools to assess surgeons' intraoperative cognitive workload. Br J Surg. 2018 Apr;105(5):491-501. doi: 10.1002/bjs.10795. Epub 2018 Feb 21. PMID 29465749
- [Background] Elhilali MM, Badaan S, Ibrahim A, Andonian S. Use of the Moses Technology to Improve Holmium Laser Lithotripsy Outcomes: A Preclinical Study. J Endourol. 2017 Jun;31(6):598-604. doi: 10.1089/end.2017.0050. Epub 2017 Apr 25. PMID 28340540
- [Background] Ibrahim A, Badaan S, Elhilali MM, Andonian S. Moses technology in a stone simulator. Can Urol Assoc J. 2018 Apr;12(4):127-130. doi: 10.5489/cuaj.4797. Epub 2017 Dec 22. PMID 29319478
- [Background] Mullerad M, Aguinaga JRA, Aro T, Kastin A, Goldin O, Kravtsov A, Assadi A, Badaan S, Amiel GE. Initial Clinical Experience with a Modulated Holmium Laser Pulse-Moses Technology: Does It Enhance Laser Lithotripsy Efficacy? Rambam Maimonides Med J. 2017 Oct 16;8(4):e0038. doi: 10.5041/RMMJ.10315. PMID 28914602
- [Background] Stern KL, Monga M. The Moses holmium system - time is money. Can J Urol. 2018 Jun;25(3):9313-9316. PMID 29900818
- [Background] Humphreys MR, Shah OD, Monga M, Chang YH, Krambeck AE, Sur RL, Miller NL, Knudsen BE, Eisner BH, Matlaga BR, Chew BH. Dusting versus Basketing during Ureteroscopy-Which Technique is More Efficacious? A Prospective Multicenter Trial from the EDGE Research Consortium. J Urol. 2018 May;199(5):1272-1276. doi: 10.1016/j.juro.2017.11.126. Epub 2017 Dec 16. PMID 29253579
- [Derived] Gelikman DG, Ibanez KR, Reed AM, Hsi RS, Nimmagadda N, Miller NL. Factors Affecting Holmium Laser Efficiency: Comparison of Laryngeal Mask Airway and Endotracheal Intubation During Ureteroscopy for Renal Stones. J Endourol. 2024 Jan;38(1):8-15. doi: 10.1089/end.2023.0294. Epub 2023 Dec 7. PMID 37933898

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moses Laser Lithotripsy | Standard Laser Lithotripsy
Started | 86 | 85
Completed | 74 | 79
Not Completed | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Laser Lithotripsy | Moses Laser Lithotripsy | Total
Number analyzed (Participants) | 79 | 74 | 153
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [48 to 72] | 61 [50 to 69] | 61 [50 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 38 | 82
  Male | 35 | 36 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 70 | 65 | 135
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Body mass index (BMI, kg/m2) [Median (Inter-Quartile Range); unit: kg/m2] | 31.14 [26.45 to 34.35] | 30.21 [25.71 to 35.70] | 30.45 [25.83 to 35.19]
Laterality of stones [Count of Participants; unit: Participants]
  Right | 35 | 35 | 70
  Left | 44 | 39 | 83
Maximum axial stone size [Median (Inter-Quartile Range); unit: millimeters] | 9.7 [8.0 to 11.5] | 10.0 [8.0 to 12.5] | 10.0 [8.0 to 12.0]

OUTCOME MEASURES:

1. Primary Outcome: Operative Time
Description: Total operative times between Moses holmium laser lithotripsy and non-Moses holmium laser lithotripsy in the ureteroscopic treatment of renal stones using a dusting technique
Time Frame: Beginning to end of procedure time, assessed up to 2 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Standard Laser Lithotripsy | Moses Laser Lithotripsy
Number analyzed (Participants) | 79 | 74
minutes | 36 [30 to 50] | 37 [31 to 51]

2. Secondary Outcome: Stone Retropulsion
Description: Stone movement during laser lithotripsy will be recorded on video and graded on a Likert scale by blinded reviewers. Video could not be taken for all trial patients. Videos were obtained and stored when feasible.
Time Frame: First 20 seconds of laser lithotripsy
Population: Video could not be taken for all trial patients. Videos were obtained and stored when feasible.
Measure: Number; unit: videos (1 video per participant)
Arm/Group | Standard Laser Lithotripsy | Moses Laser Lithotripsy
Number analyzed (Participants) | 61 | 57
videos (1 video per participant)
  No retropulsion | 18 | 27
  Some retropulsion | 32 | 21
  Significant retropulsion | 11 | 9

ADVERSE EVENTS:
Time Frame: 30 days postoperatively
Arm/Group | Standard Laser Lithotripsy | Moses Laser Lithotripsy
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/74
Serious Adverse Events (participants affected / at risk) | 7/79 | 4/74
Other Adverse Events (participants affected / at risk) | 3/79 | 3/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Laser Lithotripsy (N=79) | Moses Laser Lithotripsy (N=74)
Severe urinary tract infection (Infections and infestations) | 5 | 2 — Sepsis from urinary source, pyelonephritis
Repeat surgical intervention for pain or stone fragments (Surgical and medical procedures) | 1 | 2
Readmission for pain (Renal and urinary disorders) | 0 | 1
Urinary retention requiring foley catheter placement (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Laser Lithotripsy (N=79) | Moses Laser Lithotripsy (N=74)
Present to ED with renal colic (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 1
Presented to ED with pain, fevers and treated for UTI (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT04505956/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04505956/ICF_001.pdf